CLINICAL TRIAL: NCT05222074
Title: Venous Congestion Rather Than Intraoperative Hypotension is Associated With Acute Adverse Kidney Events After Cardiac Surgery
Brief Title: Effect of CVP and IOH on AKI and AKD
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, HONG LIANG, Doctor, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20211224-09
Record Dates: First submitted 2021-12-26; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Acute Kidney Injury; Acute Kidney Disease
Keywords: Acute kidney injury; Intraoperative hypotension; Central venous pressure; Acute kidney disease; Cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- CVP ≥ 12: central venous pressure ≥12 mmHg
  Interventions: Other: Venous congestion
- CVP ≥ 16: central venous pressure ≥16 mmHg
  Interventions: Other: Venous congestion
- CVP ≥ 20: central venous pressure ≥20 mmHg
  Interventions: Other: Venous congestion
- MAP ≤ 55 mmHg: mean arterial pressure ≤55 mmHg
  Interventions: Other: Introperation hypotension
- MAP ≤ 65 mmHg: mean arterial pressure ≤65 mmHg
  Interventions: Other: Introperation hypotension
- MAP ≤ 75 mmHg: mean arterial pressure ≤75 mmHg
  Interventions: Other: Introperation hypotension

INTERVENTIONS:
Other: Venous congestion — Venous congestion exposures were quantified as area under the curve (AUC) of central venous pressure ≥12, 16 or 20 mmHg
  Groups: CVP ≥ 12; CVP ≥ 16; CVP ≥ 20
Other: Introperation hypotension — Introperation hypotension exposures were quantified as area under the curve (AUC) of mean arterial pressure ≤55, 65, 75 mmHg
  Groups: MAP ≤ 55 mmHg; MAP ≤ 65 mmHg; MAP ≤ 75 mmHg

SUMMARY:
This study was aimed to explore the effect of intraoperative venous congestion and intraoperative hypotension (IOH) on acute adverse kidney events, defined as acute kidney injury (AKI) and acute kidney disease (AKD), after cardiac surgery

DETAILED DESCRIPTION:
Venous congestion and IOH were primary exposures and quantified as area under the curve (AUC) of central venous pressure ≥12, 16 or 20 mmHg or mean arterial pressure ≤55, 65, 75 mmHg. The primary outcome was AKI or AKD defined as renal dysfunction persisting > 7 days after surgery. Multivariable logistic regression and Cox proportional hazard models were used to determine the association between intraoperative venous congestion/hypotension and postoperative acute adverse kidney events, respectively, adjusted for relevant confounding factors and multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older,
* Patients underwent cardiac surgery (coronary artery bypass grafting, heart valve surgery, heart transplant or surgical excision of intracardiac myxoma)
* Patients receiving invasive intraoperative BP monitoring during surgery
* Patients underwent cardiopulmonary bypass (CPB) during surgery

Exclusion Criteria:

* Pre-existing renal insufficiency defined by presence of abnormal preoperative serum creatinine ≥ 133 μmol/L and/or preoperative diagnosis of renal insufficiency within 6 months'preoperative period.
* Patients with preoperative dialysis dependence within 60 days before the index surgical procedure,
* Surgical duration less than 30 minutes
* Surgery on the aorta
* Insufficient hemodynamic and laboratory data for outcomes and/or exposure ascertainment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults undergoing cardiac surgery between 2016 and 2020 (data analysed in 2021) using electronic health records collected from the Nanjing First Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5127 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
CSA-AKI | 7 days post operation
  Cardiovascular surgery associated acute kidney injury. AKI was defined using the Kidney Disease: Improving Global Outcome (KDIGO) Clinical Practice Guideline for Acute Kidney Injury as an absolute increase in serum creatinine of ≥ 26 μmol/L within 48 hours or an increase in serum creatinine beyond 1.5 times the baseline value within 7 days
AKD | 8 to 90 days post operation
  Acute Kidney Disease, which was defined according to the criteria recommended by the Acute Disease Quality Initiative (ADQI) workgroup.4 AKI was quantified within the 7 days' postoperative period, while AKD was defined as serum creatinine value elevated to 1.5 times the baseline value between 8- and 90-day post-operation period.

SECONDARY OUTCOMES:
Incidence of AKD of stage 2 and above | 8 to 90 days post operation
  incidence of AKD of stage 2 and above, defined as increase in serum creatinine beyond 2.0 times the baseline value between 8- and 90-day post-operation period.
RRT initiation | from the end of operation to the discharge from hospital, up to 90 days.
  renal replacement theray (RRT) initiation
value of eGFR | 7 days after operation
  postoperative estimated glomerular filtration rate (eGFR), which was calculated by MDRD Equation.
inpatient mortality | 30 days after inhospital
  mortality during hospital stay
ICU length of stay | from the end of operation to the discharge from ICU, up to 90 days.
  days stay in ICU
length of hospital stay | from the end of operation to the discharge from hospital, up to 90 days.
  days stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Lihai Chen, PhD, Principal Investigator — chenlihai1983@163.com
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vervoort D, Swain JD, Pezzella AT, Kpodonu J. Cardiac Surgery in Low- and Middle-Income Countries: A State-of-the-Art Review. Ann Thorac Surg. 2021 Apr;111(4):1394-1400. doi: 10.1016/j.athoracsur.2020.05.181. Epub 2020 Aug 6. PMID 32771467
- [Background] Weisse AB. Cardiac surgery: a century of progress. Tex Heart Inst J. 2011;38(5):486-90. PMID 22163121
- [Background] Wang Y, Bellomo R. Cardiac surgery-associated acute kidney injury: risk factors, pathophysiology and treatment. Nat Rev Nephrol. 2017 Nov;13(11):697-711. doi: 10.1038/nrneph.2017.119. Epub 2017 Sep 4. PMID 28869251
- [Background] Ortega-Loubon C, Fernandez-Molina M, Carrascal-Hinojal Y, Fulquet-Carreras E. Cardiac surgery-associated acute kidney injury. Ann Card Anaesth. 2016 Oct-Dec;19(4):687-698. doi: 10.4103/0971-9784.191578. PMID 27716701
- [Background] Swaminathan M, Hudson CC, Phillips-Bute BG, Patel UD, Mathew JP, Newman MF, Milano CA, Shaw AD, Stafford-Smith M. Impact of early renal recovery on survival after cardiac surgery-associated acute kidney injury. Ann Thorac Surg. 2010 Apr;89(4):1098-104. doi: 10.1016/j.athoracsur.2009.12.018. PMID 20338313
- [Background] Robert AM, Kramer RS, Dacey LJ, Charlesworth DC, Leavitt BJ, Helm RE, Hernandez F, Sardella GL, Frumiento C, Likosky DS, Brown JR; Northern New England Cardiovascular Disease Study Group. Cardiac surgery-associated acute kidney injury: a comparison of two consensus criteria. Ann Thorac Surg. 2010 Dec;90(6):1939-43. doi: 10.1016/j.athoracsur.2010.08.018. PMID 21095340
- [Background] Englberger L, Suri RM, Li Z, Casey ET, Daly RC, Dearani JA, Schaff HV. Clinical accuracy of RIFLE and Acute Kidney Injury Network (AKIN) criteria for acute kidney injury in patients undergoing cardiac surgery. Crit Care. 2011;15(1):R16. doi: 10.1186/cc9960. Epub 2011 Jan 13. PMID 21232094
- [Background] Arora P, Rajagopalam S, Ranjan R, Kolli H, Singh M, Venuto R, Lohr J. Preoperative use of angiotensin-converting enzyme inhibitors/angiotensin receptor blockers is associated with increased risk for acute kidney injury after cardiovascular surgery. Clin J Am Soc Nephrol. 2008 Sep;3(5):1266-73. doi: 10.2215/CJN.05271107. Epub 2008 Jul 30. PMID 18667735
- [Background] Ouzounian M, Buth KJ, Valeeva L, Morton CC, Hassan A, Ali IS. Impact of preoperative angiotensin-converting enzyme inhibitor use on clinical outcomes after cardiac surgery. Ann Thorac Surg. 2012 Feb;93(2):559-64. doi: 10.1016/j.athoracsur.2011.10.058. PMID 22269723
- [Background] Welten GM, Chonchol M, Schouten O, Hoeks S, Bax JJ, van Domburg RT, van Sambeek M, Poldermans D. Statin use is associated with early recovery of kidney injury after vascular surgery and improved long-term outcome. Nephrol Dial Transplant. 2008 Dec;23(12):3867-73. doi: 10.1093/ndt/gfn381. Epub 2008 Jul 15. PMID 18628367